CLINICAL TRIAL: NCT05245162
Title: Fertility Changes Due to Cancer: an Investigation of Meaning, Psychological Distress, and Psychological Support Needs of Young Women With Breast Cancer
Brief Title: Fertility Changes Due to Cancer: an Investigation of Meaning, Psychological Distress, and Psychologi
Status: Withdrawn | Type: Observational
Why Stopped: Low accrual
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 19-1812.cc
Record Dates: First submitted 2021-09-23; First posted 2022-02-17 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants: Study participants with breast cancer
- Participants partner: Study participants partner

SUMMARY:
Establish the relationship between meaning and psychological distress in young women with breast cancer who experienced reproductive concerns due to cancer diagnosis and treatment and their partners.

DETAILED DESCRIPTION:
This research will focus on identifying avenues for improving the quality of life of young women with breast cancer who endorse reproductive concerns due to cancer diagnosis and treatment, as there is an increased likelihood of distress and decreased likelihood of receiving information and appropriate psychological care. Existential distress appears to play a role in coping with infertility due to cancer (8) and thus the relationship between this distress and the other types of reproductive concerns warrants further exploration. The proposed project will use a mixed methods design to characterize the relationship between sense of meaning and purpose and psychological distress and assess psychosocial support needs of these young women. It will also assess the experience of the identified partners of these young women.

ELIGIBILITY:
Participant Inclusion Criteria:

* Provision to complete the consent form.
* Stated willingness to comply with all study procedures and be available for the duration of the study.
* Able to confirm they have a valid and private email account and access to the internet.
* Patients age 18 to 45 with a diagnosis of breast cancer. Patients will endorse that they experience reproductive concerns due to cancer as assessed by a single screening item.
* Fluent and literate in English.

Partner participant inclusion criteria:

* Provision to complete the consent form.
* Stated willingness to comply with all study procedures and be available for the duration of the study.
* Able to confirm they have a valid and private email account and access to the internet.
* Be the identified supportive partner of a study participant.
* Fluent and literate in English.

Exclusion Criteria:

* An individual who fails to meet any of the inclusion criteria will be excluded from participation in this study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Female. Ages 18 to 45. Ambulatory outpatient oncology.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-08-11 (Actual); Study Completion 2021-08-11 (Actual)

PRIMARY OUTCOMES:
Establishing distress level using questionnaires | 6 months
  Establish the relationship between meaning and psychological distress in young women with breast cancer who experienced reproductive concerns due to cancer diagnosis and treatment and their partners.

SECONDARY OUTCOMES:
Establish supports needs from established questionnaire | 6 months
  Clarify the psychosocial support needs of young women with breast cancer who experienced reproductive concerns due to cancer diagnosis and treatment and their partners

CONTACTS AND LOCATIONS:
Overall Officials: Elissa Kolva, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Health, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No